CLINICAL TRIAL: NCT06639711
Title: Taurine Affects the Progression of Senile Cataract: a Single-arm Pre-post Intervention Study
Brief Title: Taurine Eye Drops May Prevent the Progression of Cataract
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Of Anbar (Other)
Responsible Party: Principal Investigator, Atheer Zgair, Asst. Prof. Dr. Atheer Zgair, University Of Anbar
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UOANBAR-170
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Taurine

STUDY DESIGN:
Intervention Model Description: single-arm pre-post intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Application of Taurine-containing Eye Drops (Experimental)
  Interventions: Drug: Taurine

INTERVENTIONS:
Drug: Taurine — Taurine-containing eye drops (VIZILOTON) are applied 4 times daily for a period of one year
  Other Names: VIZILOTIN Eye Drops

SUMMARY:
The aim of the current intervention study is to determine the effectiveness of taurine containing eye drops (available under brand name VIZILOTON) to prevent the progression of grade I and II senile cataract.

This study could answer:

* Dose continuous use of taurine-containing eye drops could prevent further deterioration of vision in mild cases of cataract?
* The acceptance/ compliance of participants to taurine-containing eye drops.
* Could long-term use of taurine-containing eye drops cause adverse effect(s)?

Participants will:

* Take taurine-containing eye drops (VIZILOTON eye drops) 4 times a day for one year.
* Visit eye clinic every 3 months for assessment and visual examination.
* Keep notes for their symptoms and their adherence to treatment.

ELIGIBILITY:
Inclusion Criteria:

* The presence of grade I or II senile cataract on one or two eyes.

Exclusion Criteria:

* clinical signs of glaucoma
* history of amblyopia, eye surgery, argon or YAG laser eye treatment, or major eye trauma
* history of iritis, retinal crystalline deposits, or optic nerve disease
* visually significant fundus pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Visual Acuity | 1 Year

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Nahrain Eye Clinics, Ramadi, Al-Anbar Governorate, Iraq

IPD SHARING:
Plan to Share IPD: No